CLINICAL TRIAL: NCT02654990
Title: A Multicenter, Randomized, Open-label Phase 2 Study Evaluating the Safety and Efficacy of Three Different Regimens of Oral Panobinostat in Combination With Subcutaneous Bortezomib and Oral Dexamethasone in Patients With Relapsed or Relapsed/Refractory Multiple Myeloma Who Have Been Previously Exposed to Immunomodulatory Agents
Brief Title: Panobinostat/Bortezomib/Dexamethasone in Relapsed or Relapsed-and-refractory Multiple Myeloma
Acronym: PANORAMA_3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: pharmaand GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589D2222; 2015-001564-19 (EudraCT Number)
Record Dates: First submitted 2015-12-16; First posted 2016-01-13 (Estimated); Results first posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; relapsed or relapsed/refractory; LBH589; panobinostat; bortezomib; dexamethasone
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Panobinostat; Bortezomib; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A - 20 mg Panobinostat TIW (Experimental): 20 mg panobinostat TIW, 2 weeks on/1 week off in combination with subcutaneous bortezomib and per oral dexamethasone
  Interventions: Drug: Panobinostat Capsules; Drug: Bortezomib Injection; Drug: Dexamethasone tablets
- Arm B - 20 mg Panobinostat BIW (Experimental): 20 mg panobinostat BIW, 2 weeks on/1 week off in combination with subcutaneous bortezomib and per oral dexamethasone
  Interventions: Drug: Panobinostat Capsules; Drug: Bortezomib Injection; Drug: Dexamethasone tablets
- Arm C - 10 mg Panobinostat TIW (Experimental): 10 mg panobinostat TIW, 2 weeks on/1 week off in combination with subcutaneous bortezomib and per oral dexamethasone
  Interventions: Drug: Panobinostat Capsules; Drug: Bortezomib Injection; Drug: Dexamethasone tablets

INTERVENTIONS:
Drug: Panobinostat Capsules — 20 mg, 10 mg or 15 mg (for dose reductions only)
  Other Names: PAN; LBH589; Farydak
Drug: Bortezomib Injection — 1.3 mg/square meter subcutaneous administration. Cycle 1-4: 2 weeks on/1 week off, BIW for participants ≤ 75 years at time of screening; once a week for participants > 75 years. Cycle 5+: once a week for all participants.
  Other Names: BTZ; Velcade
Drug: Dexamethasone tablets — Pre and 24 hours after bortezomib administration. Participants ≤ 75 years at time of screening: 20 mg/dose participants; > 75 years: 10 mg/dose.
  Other Names: Dex; Decadron

SUMMARY:
Note: The study data was transferred to zr pharma& following the divestment of panobinostat to pharma&. Prior to study completion under the sponsorship of Secura Bio, the study was initiated and conducted in part under the sponsorship of Novartis.

The purpose of this study is to investigate the safety and efficacy of 3 different regimens of panobinostat (20 milligrams [mg] thrice a week [TIW], 20 mg twice a week [BIW], and 10 mg TIW) in combination with subcutaneous bortezomib and dexamethasone and to provide exposure, safety and efficacy data to identify the optimal regimen of panobinostat in a randomized, 3-arm parallel design. This study will also assess the impact of administering subcutaneous bortezomib (in combination with panobinostat and dexamethasone) twice weekly for 4 cycles, and then weekly starting from Cycle 5 until disease progression in participants ≤ 75 years of age. Participants > 75 years of age will receive subcutaneous bortezomib weekly for the entire treatment period (in combination with panobinostat and dexamethasone) until disease progression.

Participants will be treated until disease progression or until they discontinue earlier due to unacceptable toxicity or for other reasons.

Participants who discontinued study treatment for reasons other than disease progression will be followed for efficacy every 6 weeks.

All participants will be followed for survival until the last participant entering long-term follow-up has completed a 3-year survival follow-up or discontinued earlier.

ELIGIBILITY:
Inclusion Criteria:

* multiple myeloma per International Myeloma Working Group 2014 definition
* requiring treatment for relapsed or relapsed/refractory disease
* measurable disease based on central protein assessment
* received 1 to 4 prior lines of therapy
* prior immunomodulatory agent(s) exposure
* acceptable lab values prior to randomization

Exclusion Criteria:

* primary refractory myeloma
* refractory to bortezomib
* concomitant anti-cancer therapy (other than bortezomib/dexamethasone and bisphosphonates)
* prior treatment with pan-deacetylase inhibitors
* clinically significant, uncontrolled heart disease and/or recent cardiac event (within 6 months prior to randomization)
* unresolved diarrhea ≥ Common Terminology Criteria for adverse events grade 2 or presence of medical condition associated with chronic diarrhea (such as irritable bowel syndrome and inflammatory bowel disease)

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2016-04-27 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2022-08-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (74):
- United States (9):
  - Novartis Investigative Site, Fayetteville, Arkansas
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Fort Collins, Colorado
  - Novartis Investigative Site, Gainesville, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Lake Success, New York
  - Novartis Investigative Site, Morgantown, West Virginia
- Novartis Investigative Site, Prahran, Victoria, Australia
- Novartis Investigative Site, Hasselt, Belgium
- Brazil (3):
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, São Paulo
- Canada (2):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Kitchener, Ontario
- Czechia (2):
  - Novartis Investigative Site, Ostrava Poruba, Czech Republic
  - Novartis Investigative Site, Prague
- France (9):
  - Novartis Investigative Site, Bayonne, Bayonne Cedex
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, La Roche-sur-Yon
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Metz
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
- Germany (8):
  - Novartis Investigative Site, Bad Saarow
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leipzig
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Pátrai
- Hungary (4):
  - Novartis Investigative Site, Debrecen, HUN
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Nyíregyháza
- Italy (2):
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Rimini, RN
- Lebanon (2):
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, Sidon
- Netherlands (2):
  - VUmc, Hematology, PK2 BR012, Amsterdam
  - Albert Schweitzer ziekenhuis, Hematology, Dordrecht
- Novartis Investigative Site, Oslo, Norway
- Poland (4):
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Torun
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Portugal (2):
  - Novartis Investigative Site, Braga
  - Novartis Investigative Site, Porto
- Russia (2):
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
- South Korea (2):
  - Novartis Investigative Site, Hwasun
  - Novartis Investigative Site, Seoul
- Spain (7):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Zaragoza
- Sweden (3):
  - Novartis Investigative Site, Luleå
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Uppsala
- Thailand (3):
  - Novartis Investigative Site, Nonthaburi, Muang
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir

REFERENCES:
- [Derived] Laubach JP, Schjesvold F, Mariz M, Dimopoulos MA, Lech-Maranda E, Spicka I, Hungria VTM, Shelekhova T, Abdo A, Jacobasch L, Polprasert C, Hajek R, Illes A, Wrobel T, Sureda A, Beksac M, Goncalves IZ, Blade J, Rajkumar SV, Chari A, Lonial S, Spencer A, Maison-Blanche P, Moreau P, San-Miguel JF, Richardson PG. Efficacy and safety of oral panobinostat plus subcutaneous bortezomib and oral dexamethasone in patients with relapsed or relapsed and refractory multiple myeloma (PANORAMA 3): an open-label, randomised, phase 2 study. Lancet Oncol. 2021 Jan;22(1):142-154. doi: 10.1016/S1470-2045(20)30680-X. Epub 2020 Dec 7. PMID 33301738

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A - Panobinostat (20 mg, TIW): Participants received 20 milligrams (mg) panobinostat thrice a week (TIW), 2 weeks on/1 week off in combination with subcutaneous bortezomib and oral dexamethasone.
- Arm B - Panobinostat (20 mg, BIW): Participants received 20 mg panobinostat twice a week (BIW), 2 weeks on/1 week off in combination with subcutaneous bortezomib and oral dexamethasone.
- Arm C - Panobinostat (10 mg, TIW): Participants received 10 mg panobinostat TIW, 2 weeks on/1 week off in combination with subcutaneous bortezomib and oral dexamethasone.
Period: Overall Study
Arm/Group | Arm A - Panobinostat (20 mg, TIW) | Arm B - Panobinostat (20 mg, BIW) | Arm C - Panobinostat (10 mg, TIW)
Started (Full analysis set (FAS): all participants to whom study treatment was assigned by randomization.) | 82 | 83 | 83
Received at Least 1 Dose of Study Drug (Safety Set: all participants who received any study treatment.) | 79 | 82 | 80
Completed | 82 | 83 | 83
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): all participants to whom study treatment was assigned by randomization.
Groups:
- Arm A - Panobinostat (20 mg, TIW): Participants received 20 mg panobinostat TIW, 2 weeks on/1 week off in combination with subcutaneous bortezomib and oral dexamethasone.
- Arm B - Panobinostat (20 mg, BIW): Participants received 20 mg panobinostat BIW, 2 weeks on/1 week off in combination with subcutaneous bortezomib and oral dexamethasone.
- Total: Total of all reporting groups
Arm/Group | Arm A - Panobinostat (20 mg, TIW) | Arm B - Panobinostat (20 mg, BIW) | Arm C - Panobinostat (10 mg, TIW) | Total
Number analyzed (Participants) | 82 | 83 | 83 | 248
Age, Continuous [Median (Full Range); unit: years] | 67.0 [45 to 83] | 65.0 [47 to 87] | 66.0 [33 to 84] | 66.5 [33 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 39 | 33 | 112
  Male | 42 | 44 | 50 | 136
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not Hispanic or Latino | 49 | 43 | 38 | 130
  Ethnicity: Southeast Asian | 4 | 4 | 6 | 14
  Ethnicity: Hispanic or Latino | 4 | 5 | 9 | 18
  Ethnicity: Other | 17 | 23 | 26 | 66
  Ethnicity: Unknown/Not Reported | 8 | 8 | 4 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 73 | 72 | 68 | 213
  Race: Asian | 6 | 7 | 10 | 23
  Race: Black or African American | 1 | 0 | 2 | 3
  Race: Other | 2 | 4 | 3 | 9
Eastern Cooperative Oncology Group Performance Status [Count of Participants; unit: Participants] — Scale to assess disease progression and disease effects on daily living abilities, as well as determine appropriate treatment and prognosis. Status range includes: 0 (fully active); 1 (restricted physical activity); 2 (unable to carry out work activities); 3 (limited self-care); 4 (completely disabled).
  Participants
    0 | 38 | 38 | 42 | 118
    1 | 36 | 45 | 35 | 116
    2 | 8 | 0 | 6 | 14
    3 | 0 | 0 | 0 | 0
    4 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a confirmed partial response (PR) or better (immunophenotypic complete response [iCR] or stringent complete response [sCR] or complete response [CR] or very good partial response [VGPR]) as their best overall response after completion of up to 8 cycles of assigned study regimen. Each cycle was 21 days long. Best overall response was the best post-baseline confirmed overall response observed in a given participant and was determined based on overall responses observed at all post-baseline response assessments, recorded from randomization until progressive disease (PD), death, start of new therapy, withdrawal of consent, or end of study, whatever came first. ORR was assessed blindly per independent review committee (IRC) according to International Myeloma Working Group (IMWG) criteria.
Time Frame: Up to 168 days
Population: Full analysis set (FAS): all participants to whom study treatment was assigned by randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A - Panobinostat (20 mg, TIW) | Arm B - Panobinostat (20 mg, BIW) | Arm C - Panobinostat (10 mg, TIW)
Number analyzed (Participants) | 82 | 83 | 83
percentage of participants | 62.2 [50.8 to 72.7] | 65.1 [53.8 to 75.2] | 50.6 [39.4 to 61.8]

2. Secondary Outcome: ORR Throughout the Study
Description: ORR is defined as the percentage of participants with a confirmed PR or better (iCR or sCR or CR or VGPR) as their best overall response throughout the entire study. Best overall response was the best post-baseline confirmed overall response observed in a given participant and was determined based on overall responses observed at all post-baseline response assessments, recorded from randomization until PD, death, start of new therapy, withdrawal of consent or end of study, whatever came first. ORR was assessed blindly per IRC according to IMWG criteria.
Time Frame: Up to 5.2 years
Population: Full analysis set (FAS): all participants to whom study treatment was assigned by randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A - Panobinostat (20 mg, TIW) | Arm B - Panobinostat (20 mg, BIW) | Arm C - Panobinostat (10 mg, TIW)
Number analyzed (Participants) | 82 | 83 | 83
percentage of participants | 62.2 [50.8 to 72.7] | 67.5 [56.3 to 77.4] | 53.0 [41.7 to 64.1]

3. Secondary Outcome: iCR Rate
Description: iCR, based on IMWG criteria per blinded IRC assessment, is defined as: negative immunofixation of serum and urine; disappearance of any soft tissue plasmacytoma(s), in the case of any presence of soft tissue plasmacytoma(s) at baseline; less than 5% plasma cells in bone marrow; normal free light chain (FLC) ratio; absence of clonal plasma cells in bone marrow analyzed by immunohistochemistry or 2- to 4-color flow cytometry; absence of phenotypically aberrant plasma cells (clonal) in bone marrow (BM) with a minimum of 1 million total BM cells analyzed by multiparametric flow cytometry (>4 colors). Results reported as percentage of participants achieving iCR.
Time Frame: Up to 5.2 years
Population: Full analysis set (FAS): all participants to whom study treatment was assigned by randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A - Panobinostat (20 mg, TIW) | Arm B - Panobinostat (20 mg, BIW) | Arm C - Panobinostat (10 mg, TIW)
Number analyzed (Participants) | 82 | 83 | 83
percentage of participants | 3.7 | 1.2 | 1.2

4. Secondary Outcome: sCR Rate
Description: sCR, based on IMWG criteria per blinded IRC assessment, is defined as: negative immunofixation of serum and urine; disappearance of any soft tissue plasmacytoma(s), in the case of any presence of soft tissue plasmacytoma(s) at baseline; less than 5% plasma cells in bone marrow; normal FLC ratio; absence of clonal plasma cells in bone marrow analyzed by immunohistochemistry or 2- to 4-color flow cytometry. Results reported as percentage of participants achieving sCR.
Time Frame: Up to 5.2 years
Population: Full analysis set (FAS): all participants to whom study treatment was assigned by randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A - Panobinostat (20 mg, TIW) | Arm B - Panobinostat (20 mg, BIW) | Arm C - Panobinostat (10 mg, TIW)
Number analyzed (Participants) | 82 | 83 | 83
percentage of participants | 1.2 | 1.2 | 3.6

5. Secondary Outcome: CR Rate
Description: CR, based on IMWG criteria per blinded IRC assessment, is defined as: negative immunofixation of serum and urine; disappearance of any soft tissue plasmacytoma(s), in the case of any presence of soft tissue plasmacytoma(s) at baseline; less than 5% plasma cells in bone marrow; in case the only measurable disease at baseline is the serum FLC assessment, a normal FLC ratio of 0.26 to 1.65 is required additionally to qualify for CR. Results reported as percentage of participants achieving CR.
Time Frame: Up to 5.2 years
Population: Full analysis set (FAS): all participants to whom study treatment was assigned by randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A - Panobinostat (20 mg, TIW) | Arm B - Panobinostat (20 mg, BIW) | Arm C - Panobinostat (10 mg, TIW)
Number analyzed (Participants) | 82 | 83 | 83
percentage of participants | 8.5 | 8.4 | 2.4

6. Secondary Outcome: VGPR Rate
Description: VGPR, based on IMWG criteria per blinded IRC assessment, is defined as: serum and/or urine M protein detectable by immunofixation but not on protein electrophoresis, or ≥90% reduction from baseline in serum) and urine M protein <100 milligrams/24 hours); in the case of the presence of any soft tissue plasmacytoma(s) at baseline, a reduction in the sum of the products of the cross-diameters by ≥50% from baseline is required; in case the only measurable disease in a participant at baseline is the serum FLC level (that is, no measurable disease in serum and urine PEP), a decrease of >90% in the difference between involved and uninvolved FLC levels from baseline is required. Results reported as percentage of participants achieving VGPR.
Time Frame: Up to 5.2 years
Population: Full analysis set (FAS): all participants to whom study treatment was assigned by randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A - Panobinostat (20 mg, TIW) | Arm B - Panobinostat (20 mg, BIW) | Arm C - Panobinostat (10 mg, TIW)
Number analyzed (Participants) | 82 | 83 | 83
percentage of participants | 19.5 | 25.3 | 20.5

7. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS, assessed based on IMWG criteria per blind IRC assessment, is defined as the time from date of randomization to date of first documented disease progression or death (regardless of cause of death).
Time Frame: Up to 5.2 years
Population: Full analysis set (FAS): all participants to whom study treatment was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A - Panobinostat (20 mg, TIW) | Arm B - Panobinostat (20 mg, BIW) | Arm C - Panobinostat (10 mg, TIW)
Number analyzed (Participants) | 82 | 83 | 83
months | 15 [7.4 to 24.7] | 13 [7.0 to 13.8] | 8 [5.0 to 10.7]

8. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from date of randomization to the date of death due to any cause.
Time Frame: Up to 5.2 years
Population: Full analysis set (FAS): all participants to whom study treatment was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A - Panobinostat (20 mg, TIW) | Arm B - Panobinostat (20 mg, BIW) | Arm C - Panobinostat (10 mg, TIW)
Number analyzed (Participants) | 82 | 83 | 83
months | 35 [27.8 to NA] — Not evaluable due to insufficient number of events | 32 [30.7 to NA] — Not evaluable due to insufficient number of events | 22 [18.6 to NA] — Not evaluable due to insufficient number of events

9. Secondary Outcome: Maximum Plasma Concentration (Cmax): Panobinostat
Description: Serial blood samples were collected for panobinostat Cmax analysis. Results are reported in nanograms/milliliter (ng/mL).
Time Frame: Cycle 1 Day 1 (Pre-dose, up to 8 hours post dose)
Population: Pharmacokinetics Analysis Set (PAS): all participants with at least 1 evaluable pharmacokinetics concentration of panobinostat after dosing on Day 1. Here, 'Overall Number of Participants Analyzed' refers to the number of evaluable participants analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm A - Panobinostat (20 mg, TIW) | Arm B - Panobinostat (20 mg, BIW) | Arm C - Panobinostat (10 mg, TIW)
Number analyzed (Participants) | 50 | 64 | 62
ng/mL | 14.30 (7.77) | 14.12 (8.96) | 6.13 (3.51)

10. Secondary Outcome: Cmax: Bortezomib
Description: Serial blood samples were collected for bortezomib Cmax analysis. Results are reported in ng/mL.
Time Frame: Cycle 1 Day 1 (Pre-dose, up to 8 hours post dose)
Population: Pharmacokinetics Analysis Set (PAS): all participants with at least 1 evaluable pharmacokinetics concentration of bortezomib after dosing on Day 1. Here, 'Overall Number of Participants Analyzed' refers to the number of evaluable participants analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm A - Panobinostat (20 mg, TIW) | Arm B - Panobinostat (20 mg, BIW) | Arm C - Panobinostat (10 mg, TIW)
Number analyzed (Participants) | 61 | 69 | 63
ng/mL | 16.67 (7.79) | 19.47 (10.00) | 18.29 (8.80)

11. Secondary Outcome: Time to Reach Cmax (Tmax): Panobinostat
Description: Serial blood samples were collected for panobinostat Tmax analysis. Results are reported in hours.
Time Frame: Cycle 1 Day 1 (Pre-dose, up to 8 hours post dose)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Arm A - Panobinostat (20 mg, TIW) | Arm B - Panobinostat (20 mg, BIW) | Arm C - Panobinostat (10 mg, TIW)
Number analyzed (Participants) | 50 | 64 | 62
hours | 1.93 (1.53) | 1.80 (1.63) | 1.82 (1.53)

12. Secondary Outcome: Tmax: Bortezomib
Description: Serial blood samples were collected for bortezomib Tmax analysis. Results are reported in hours.
Time Frame: Cycle 1 Day 1 (Pre-dose, up to 8 hours post dose)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Arm A - Panobinostat (20 mg, TIW) | Arm B - Panobinostat (20 mg, BIW) | Arm C - Panobinostat (10 mg, TIW)
Number analyzed (Participants) | 61 | 69 | 63
hours | 0.84 (0.46) | 0.77 (0.36) | 0.77 (0.39)

13. Secondary Outcome: Exposure Response: Cmax for Panobinostat
Description: The exposure-response relationship was assessed utilizing Cmax (Cycle 1 Day 1) for panobinostat versus the outcomes of ORR, grade 3/4 thrombocytopenia, and grade 3/4 diarrhea. Two statistical models were used: logistic regression models, in which these 3 outcomes were treated in a binary fashion according to their occurrence; Cox regression models, with the relevant outcomes being the time to occurrence of grade 3/4 thrombocytopenia and the time to occurrence of grade 3/4 diarrhea. Results are reported as model-based probability. An increase in the model-based probability indicates an increase in the occurrence of the outcomes (ORR, grade 3/4 thrombocytopenia, 3/4 diarrhea) with increasing values of Cmax (that is, with increasing dose of panobinostat).
Time Frame: Up to 5.2 Years
Population: Full analysis set (FAS): all participants to whom study treatment was assigned by randomization. Here, 'Overall Number of Participants Analyzed' refers to the number of evaluable participants analyzed.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Arm A - Panobinostat (20 mg, TIW) | Arm B - Panobinostat (20 mg, BIW) | Arm C - Panobinostat (10 mg, TIW)
Number analyzed (Participants) | 18 | 20 | 18
percent probability
  ORR by IRC (up to 8 cycles): number analyzed (Participants) | 18 | 19 | 17
  ORR by IRC (up to 8 cycles) | 63.1 [46.7 to 76.9] | 62.2 [47.5 to 75.0] | 35.3 [20.6 to 53.4]
  Grade 3/4 Thrombocytopenia: number analyzed (Participants) | 18 | 20 | 17
  Grade 3/4 Thrombocytopenia | 32.2 [17.7 to 51.2] | 28.7 [17.5 to 43.4] | 21.7 [10.6 to 39.4]
  Grade 3/4 Diarrhea | 6.2 [2.1 to 16.7] | 7.5 [3.1 to 17.2] | 2.5 [0.3 to 16.3]

14. Secondary Outcome: Change From Baseline in European Organization of Research and Treatment of Cancer (EORTC) Quality of Life Core 30-item Questionnaire (QLQ-C30) Global Health Status (GHS) Score
Description: Health-related quality of life (HRQoL) was assessed by the EORTC QLQ-C30, which is frequently employed in clinical oncology trials and is recognized as reliable and valid. The EORTC QLQ-C30 measures functional dimensions (physical, role, emotional, cognitive, and social), 3 symptom items (fatigue, nausea/vomiting, and pain), 6 single items (dyspnea, sleep disturbance, appetite loss, constipation, diarrhea and financial impact), and a global health scale (GHS) and quality-of-life scale. For each domain and item, a linear transformation is applied to standardize the score between 0 and 100. Results are presented specifically for the GHS score. A higher GHS score indicates a higher HRQoL. Each cycle was 21 days long.
Time Frame: Cycle 15 Day 1, at approximately 295 days
Population: Full analysis set (FAS): all participants to whom study treatment was assigned by randomization and who had a valid baseline HRQoL assessment and at least 1 post-baseline assessment. Here, 'Overall Number of Participants Analyzed' refers to the number of evaluable participants analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A - Panobinostat (20 mg, TIW) | Arm B - Panobinostat (20 mg, BIW) | Arm C - Panobinostat (10 mg, TIW)
Number analyzed (Participants) | 18 | 16 | 18
score on a scale | 6.0 (23.01) | 0.0 (30.12) | -4.6 (24.12)

15. Secondary Outcome: Change From Baseline in the Functional Assessment of Cancer Therapy (FACT)/Gynecologic Oncology Group-Neurotoxicity (GOG-Ntx) Neurotoxicity Subscale Score
Description: HRQoL was assessed by the FACT/GOG-Ntx, a 38-item questionnaire designed to assess general quality of life and severity and impact of neurotoxicity from systemic chemotherapy. It is frequently employed in clinical oncology trials and is recognized as a reliable and valid measure to assess symptoms associated with neurotoxicity. It focuses on 4 general quality of life domains for physical well-being, functional well-being, social/family well-being, and emotional well-being, and includes the neurotoxicity subscale domain to characterize treatment-related neurotoxicity. Results are presented specifically for the 11-item neurotoxicity subscale, which uses a 5-point rating scale (0=not at all; 1=a little bit; 2=somewhat; 3=quite a bit; 4=very much). Each item is scored from 0-4, with the severity of neurotoxicity measured as the sum of the 11 items, ranging from 0 to 44. Lower scores indicate lower neurotoxicity and higher HRQoL. Each cycle was 21 days long.
Time Frame: Cycle 15 Day 1, at approximately 295 days
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A - Panobinostat (20 mg, TIW) | Arm B - Panobinostat (20 mg, BIW) | Arm C - Panobinostat (10 mg, TIW)
Number analyzed (Participants) | 18 | 15 | 18
score on a scale | -3.6 (7.39) | -3.9 (4.19) | -0.1 (5.71)

16. Secondary Outcome: Time to Progression (TTP)
Description: TTP, based on IMWG criteria per blinded IRC assessment, is defined as the time from the date of randomization to the date of the first documented disease progression or death due to multiple myeloma.
Time Frame: Up to 5.2 years
Population: Full analysis set (FAS): all participants to whom study treatment was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A - Panobinostat (20 mg, TIW) | Arm B - Panobinostat (20 mg, BIW) | Arm C - Panobinostat (10 mg, TIW)
Number analyzed (Participants) | 82 | 83 | 83
months | 17 [8.3 to NA] — Not evaluable due to insufficient number of events | 13 [7.0 to 16.1] | 8 [5.9 to 11.6]

17. Secondary Outcome: Time to Response (TTR)
Description: TTR, based on IMWG criteria per blinded IRC assessment, is the time between date of randomization to the date of first onset of PR or better response (iCR or sCR or CR or VGPR).
Time Frame: Up to 5.2 years
Population: Full analysis set (FAS): all participants to whom study treatment was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A - Panobinostat (20 mg, TIW) | Arm B - Panobinostat (20 mg, BIW) | Arm C - Panobinostat (10 mg, TIW)
Number analyzed (Participants) | 82 | 83 | 83
months | 3 [1 to NA] — Not evaluable due to insufficient number of events | 3 [1 to NA] — Not evaluable due to insufficient number of events | 3 [1 to NA] — Not evaluable due to insufficient number of events

18. Secondary Outcome: Duration of Response (DOR)
Description: DOR, based on IMWG criteria per blinded IRC assessment, is defined as the duration from the first documented onset of PR or better (iCR or sCR or CR or VGPR) to the date of first documented disease progression or death due to multiple myeloma.
Time Frame: Up to 5.2 years
Population: Full analysis set (FAS): all participants to whom study treatment was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A - Panobinostat (20 mg, TIW) | Arm B - Panobinostat (20 mg, BIW) | Arm C - Panobinostat (10 mg, TIW)
Number analyzed (Participants) | 82 | 83 | 83
months | 22 [13.9 to NA] — Not evaluable due to insufficient number of events | 12 [8.8 to 21.3] | 10.429 [6.2 to 14.5]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed for 3 years. All-Cause Mortality was assessed from date of randomization until death, assessed up to 5.2 years.
Description: Safety Set: all participants who received any study treatment.
Arm/Group | Arm A - Panobinostat (20 mg, TIW) | Arm B - Panobinostat (20 mg, BIW) | Arm C - Panobinostat (10 mg, TIW)
All-Cause Mortality (participants affected / at risk) | 34/78 | 41/83 | 47/80
Serious Adverse Events (participants affected / at risk) | 44/78 | 40/83 | 36/80
Other Adverse Events (participants affected / at risk) | 78/78 | 82/83 | 78/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Arm A - Panobinostat (20 mg, TIW) (N=78) | Arm B - Panobinostat (20 mg, BIW) (N=83) | Arm C - Panobinostat (10 mg, TIW) (N=80)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Bicytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Methaemoglobinaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 1 | 1
Atrial Flutter (Cardiac disorders) | 1 | 0 | 0
Cardiac Failure (Cardiac disorders) | 1 | 0 | 2
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 1
Cardiac Failure Acute (Cardiac disorders) | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal Motility Disorder (Gastrointestinal disorders) | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Asthenia (General disorders) | 2 | 0 | 1
Fatigue (General disorders) | 2 | 2 | 0
Drug Withdrawal Syndrome (General disorders) | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 1
General Physical Health Deterioration (General disorders) | 0 | 3 | 0
Pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 4 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 8 | 11 | 9
Lower Respiratory Tract Infection (Infections and infestations) | 3 | 0 | 1
Bacterial Pyelonephritis (Infections and infestations) | 1 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 2 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Infection (Infections and infestations) | 1 | 0 | 1
Meningitis (Infections and infestations) | 1 | 0 | 0
Pneumonia Parainfluenza Viral (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 1 | 4 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 1 | 0
Abscess Limb (Infections and infestations) | 0 | 0 | 1
Bacterial Sepsis (Infections and infestations) | 0 | 0 | 1
Diarrhoea Infectious (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 1
Haemophilus Sepsis (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 2 | 1
Parainfluenza Virus Infection (Infections and infestations) | 0 | 1 | 0
Pneumonia Haemophilus (Infections and infestations) | 0 | 1 | 0
Pneumonia Viral (Infections and infestations) | 0 | 1 | 0
Pyelonephritis Acute (Infections and infestations) | 0 | 0 | 1
Rhinovirus Infection (Infections and infestations) | 0 | 1 | 0
Septic Shock (Infections and infestations) | 0 | 2 | 1
Streptococcal Sepsis (Infections and infestations) | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 2
Forearm Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Transfusion-related Acute Lung Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Troponin Increased (Investigations) | 1 | 1 | 0
Blood Creatine Increased (Investigations) | 0 | 1 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 0 | 1
Myocardial Necrosis Marker Increased (Investigations) | 0 | 0 | 1
Platelet Count Decreased (Investigations) | 0 | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Gastrointestinal Tract Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Haematological Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 1 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 0 | 1
Confusional State (Psychiatric disorders) | 0 | 0 | 1
Hypomania (Psychiatric disorders) | 0 | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 1 | 2
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0/39 | 1/44 | 0/48 — This adverse event only affected male participants.
Orchitis Noninfective (Reproductive system and breast disorders) | 0/39 | 1/44 | 0/48 — This adverse event only affected male participants.
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Circulatory Collapse (Vascular disorders) | 1 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Peripheral Ischaemia (Vascular disorders) | 1 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 2
Respiratory Tract Infection (Infections and infestations) | 3 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4.9% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A - Panobinostat (20 mg, TIW) (N=78) | Arm B - Panobinostat (20 mg, BIW) (N=83) | Arm C - Panobinostat (10 mg, TIW) (N=80)
Thrombocytopenia (Blood and lymphatic system disorders) | 43 | 37 | 26
Anaemia (Blood and lymphatic system disorders) | 33 | 22 | 24
Neutropenia (Blood and lymphatic system disorders) | 25 | 16 | 10
Leukopenia (Blood and lymphatic system disorders) | 5 | 1 | 2
Cataract (Eye disorders) | 6 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 51 | 53 | 39
Nausea (Gastrointestinal disorders) | 29 | 29 | 13
Constipation (Gastrointestinal disorders) | 21 | 16 | 18
Vomiting (Gastrointestinal disorders) | 16 | 21 | 6
Abdominal Pain Upper (Gastrointestinal disorders) | 12 | 9 | 1
Dyspepsia (Gastrointestinal disorders) | 9 | 3 | 4
Abdominal Pain (Gastrointestinal disorders) | 5 | 11 | 7
Flatulence (Gastrointestinal disorders) | 4 | 2 | 1
Fatigue (General disorders) | 27 | 25 | 24
Asthenia (General disorders) | 25 | 29 | 15
Oedema Peripheral (General disorders) | 23 | 14 | 14
Pyrexia (General disorders) | 10 | 12 | 10
Non-cardiac Chest Pain (General disorders) | 4 | 3 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 20 | 12 | 21
Respiratory Tract Infection (Infections and infestations) | 13 | 8 | 8
Urinary Tract Infection (Infections and infestations) | 11 | 8 | 2
Bronchitis (Infections and infestations) | 9 | 8 | 1
Conjunctivitis (Infections and infestations) | 5 | 4 | 1
Respiratory Tract Infection Viral (Infections and infestations) | 4 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 4
Nasopharyngitis (Infections and infestations) | 2 | 6 | 8
Pneumonia (Infections and infestations) | 2 | 5 | 4
Influenza (Infections and infestations) | 1 | 4 | 6
Platelet Count Decreased (Investigations) | 11 | 9 | 5
Blood Creatinine Increased (Investigations) | 9 | 7 | 4
Alanine Aminotransferase Increased (Investigations) | 8 | 2 | 2
C-Reactive Protein Increased (Investigations) | 4 | 3 | 1
Neutrophil Count Decreased (Investigations) | 4 | 0 | 2
White Blood Cell Count Decreased (Investigations) | 4 | 0 | 0
Weight Decreased (Investigations) | 6 | 5 | 3
Aspartate Aminotransferase Increased (Investigations) | 5 | 2 | 0
Weight Increased (Investigations) | 2 | 6 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 14 | 9 | 7
Decreased Appetite (Metabolism and nutrition disorders) | 13 | 16 | 10
Hypocalcaemia (Metabolism and nutrition disorders) | 7 | 3 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 6 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 7 | 3
Dehydration (Metabolism and nutrition disorders) | 3 | 2 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 8 | 10
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 9 | 4 | 7
Bone Pain (Musculoskeletal and connective tissue disorders) | 5 | 5 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 5 | 6 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 11 | 5
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2 | 6 | 5
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 5
Neuropathy Peripheral (Nervous system disorders) | 20 | 22 | 14
Peripheral Sensory Neuropathy (Nervous system disorders) | 16 | 9 | 11
Dizziness (Nervous system disorders) | 13 | 12 | 5
Headache (Nervous system disorders) | 7 | 6 | 3
Paraesthesia (Nervous system disorders) | 4 | 5 | 4
Polyneuropathy (Nervous system disorders) | 3 | 5 | 5
Dysgeusia (Nervous system disorders) | 1 | 2 | 4
Neuralgia (Nervous system disorders) | 0 | 6 | 0
Insomnia (Psychiatric disorders) | 7 | 20 | 11
Depression (Psychiatric disorders) | 4 | 1 | 3
Renal Failure (Renal and urinary disorders) | 0 | 0 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 13 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 8 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 2
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 6 | 3
Hypotension (Vascular disorders) | 7 | 6 | 1
Hypertension (Vascular disorders) | 6 | 4 | 5
Orthostatic Hypotension (Vascular disorders) | 0 | 1 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor's agreements with investigators require proposed public disclosures of trial results to be submitted to Sponsor for review prior to publication. Sponsor may request deletion of confidential information or a delay in publication to address intellectual property concerns, but Sponsor may not suppress publication of the trial results indefinitely. Sponsor may request delay of a single-center publication until after the release of a multi-site publication or an agreed upon period of time.

DOCUMENTS (2):
  • Study Protocol (2019-10-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT02654990/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT02654990/SAP_001.pdf